CLINICAL TRIAL: NCT06175286
Title: Effect of a Respiratory Training Program on Woodwind and Brass Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, MARIO ALEXANDRE GONÇALVES LOPES, Adjunct Professor, Aveiro University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Musician respiratory training
Record Dates: First submitted 2023-11-24; First posted 2023-12-18 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Respiratory Function
Keywords: Inspiratory muscle training; lung capacity; musicians
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POWERBreath (Experimental): Subjects will train with the POWERBreath twice per day, for 30 continous breaths
  Interventions: Other: POWERBreath Plus Medium Resistance training device
- Control (No Intervention): Subjects will carry on with their normal daily life

INTERVENTIONS:
Other: POWERBreath Plus Medium Resistance training device — 30 inspirations with the POWERBreath Plus Medium Resistance training device, twice per day for 5 weeks
  Arms: POWERBreath

SUMMARY:
This project will study the effect of a respiratory training program on woodwind and brass players, using an inspiratory muscle training equipment. The goal is to understand whether it is possible to develop the inspiratory muscles of wind players through regular and planned training. Fourteen young wind players will be selected, in which 7 will be male and 7 will be female, playing different instruments. Inspiratory muscle training will be performed with the POWERBreath Plus Medium Resistance, and will consist of 30 maximal inspirations, twice a day, for 5 weeks.

DETAILED DESCRIPTION:
This project will study the effect of a respiratory training program on woodwind and brass players, using an inspiratory muscle training equipment. The goal is to understand whether it is possible to develop the inspiratory muscles of wind players through regular and planned training. Fourteen young wind players will be selected, in which 7 will be male and 7 will be female, playing different instruments: transverse flute (1), oboe (2), saxophone (4), horn (4), trumpet (1), trombone (1) and tuba (1). Inspiratory muscle training will be performed with the POWERBreath Plus Medium Resistance, and will consist of 30 maximal inspirations, twice a day, for 5 weeks. The participants will be instructed on the use, handling and cleaning of the equipment. The participants will be instructed to use the equipment in a comfortable position, with a good posture, and will be instructed on how they should execute the inspiratory training: inhale to the maximum limit, with intensity, and exhale slowly and relaxed. An explanation will also be given about the calibration of the POWERbreathe, and the initial resistance level will be established based on the calculation of 50% of the Maximal Inspiratory Pressure of each participant, previously measured. Participants will also be instructed on how to increase the resistance level of POWERbreathe. The increase would be 1/4 of a level, whenever they no longer feel tired after a 30-inhalation workout. A questionnaire will be applied before, during and after the inspiratory training and they will be asked to record the daily use of the equipment in an online form, created for the purpose of recording its use by each participant. Assessment will be executed with the standard Borg Scale and the modified Borg scale. Surface electromyography (sEMG) of the right sternocleidomastoid, the right scalene muscles, the diaphragm and the right rectus abdominis will also be tested. Maximal inspiratory pressure and spirometry testing, specifically volume of forced vital capacity (FVC) or forced expiratory volume in one second (FEV1) and FEV1/FVC ratio will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or over
* 10 years of musical experience

Exclusion Criteria:

* lung disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
maximum inspiratory pressure | 5 weeks
  Maximal inspiratory pressure (MIP) is an important and non-invasive index of diaphragm strength and an independent predictor of all-cause mortality (units of measure: (cmH2O).
subjective physical effort | 5 weeks
  subjective physical effort, assessed with the Borg scale (scale: 6-20; 6= "Very, very light"; 20= "Very, very hard")
dyspnea | 5 weeks
  subjective respiratory effort, assessed with the modified Borg scale (scale: 0-10; 0= "Nothing at all"; 10= "Very, very strong")
surface electromyography (sEMG) | 5 weeks
  sEMG od the scalene, sternocleidomastoid, diaphragm and abdominal muscle activity (units of measure: millivolts)
spirometry: Forced expiratory volume in one second (VEF1) | 5 weeks
  to assess lung function: the assessment of the forced expiratory volume in the fisrt second of the expiratory effort (units of measure: milliliters)
spirometry: volume of forced vital capacity (FVC) | 5 weeks
  to assess lung function: the assessment of the total forced vital capacity (units of measure: milliliters)
spirometry: ratio between VEF1 and FVC | 5 weeks
  the ratio of the forced expiratory volume in the first one second to the forced vital capacity of the lungs. The normal value for this ratio is above 0.75-85 %, though this is age dependent (units of measure: %).

CONTACTS AND LOCATIONS:
Overall Officials: Catarina Monteiro, Principal Investigator — University of Aveiro
Locations (1):
- Escola Superior de Saúde da Universidade de Aveiro, Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: No
Data will be shared upon fundamented request.

REFERENCES:
- [Background] Drinkwater EJ, Klopper CJ. Quantifying the physical demands of a musical performance and their effects on performance quality. Med Probl Perform Art. 2010 Jun;25(2):66-71. PMID 20795334
- [Result] Arend M, Kivastik J, Maestu J. Maximal inspiratory pressure is influenced by intensity of the warm-up protocol. Respir Physiol Neurobiol. 2016 Aug;230:11-5. doi: 10.1016/j.resp.2016.05.002. Epub 2016 May 12. PMID 27181328